CLINICAL TRIAL: NCT03131180
Title: Randomized Controlled Trial: Rapid Learning Healthcare System in Pediatric Surgery
Brief Title: Rapid Learning Healthcare System in Pediatric Surgery
Acronym: RLHS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Katherine Deans (Other)
Collaborators: Society of University Surgeons (Other)
Responsible Party: Sponsor-Investigator, Katherine Deans, Director, Center for Surgical Outcomes Research, Nationwide Children's Hospital; Assistant Professor of Surgery, The Ohio State University, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB16-00537
Record Dates: First submitted 2017-04-19; First posted 2017-04-27 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Colorectal Disorders

STUDY DESIGN:
Intervention Model Description: This trial is a single center randomized controlled trial to investigate the ability of the RLHS to improve patient-centered outcomes in pediatric patients with complex colorectal diseases. Patients and caregivers are randomized to either receive access to a website that displays the colorectal RLHS dashboard prior to standard consultation or to standard consultation alone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RLHS dashboard (Experimental): Patients randomized to RLHS website access are given instructions on how the RLHS dashboard works both by phone and by email and are given open access to the RLHS dashboard website immediately after enrollment and before meeting with the CCPR clinical team for their consultation. Each user has an access code, which allows them to track their access. They maintain access to the website throughout their care in the CCPR. Patients in the RLHS access group complete the System Usability Scale (SUS; a 10 item questionnaire to evaluate software, websites, and applications) after use of the RLHS at consultation. Those in the RLHS access group also complete a 7-item exit interview either via phone or on REDCap.
  Interventions: Other: Rapid Learning Healthcare System
- Standard consultation alone (No Intervention): Those not randomized to RLHS access undergo standard consultation only.

INTERVENTIONS:
Other: Rapid Learning Healthcare System — The investigators created a Rapid Learning Healthcare System that integrates pre-specified data elements and validated surveys within the clinical workflow in order to operationalize automated research data collection and integrate predictive analytics into the electronic health record (EHR). Patients, caregivers, and physicians access data in order to make informed, shared decisions about care and align expectations about outcomes.
  Other Names: Interactive Patient Education Dashboard
  Arms: RLHS dashboard

SUMMARY:
Engaging patients and families to take an active role in their healthcare leads to improved outcomes. Providing physicians and families with near real-time data on outcomes in children with similar medical conditions can allow families to form realistic expectations and take an active role in their child's health. It also provides physicians with near real-time feedback on patient-reported outcome measures to guide both conversations and recommendations for therapy at the point-of-care.

A rapid learning healthcare system (RLHS) is a system that merges clinical research and clinical care. It is designed to collect data during routine patient care and then utilize the data to rapidly generate evidence to improve patient care, provide information to patients and families, and track quality measures.

The investigators created a RLHS that integrates pre-specified data elements and validated surveys within the clinical workflow in order to operationalize automated research data collection and integrate predictive analytics into the electronic health record (EHR). Patients, caregivers, and physicians can access data in order to make informed, shared decisions about care and align expectations about outcomes.

DETAILED DESCRIPTION:
Functional disabilities such as functional constipation, and congenital anomalies such as anorectal malformations (ARM) and Hirschsprung disease (HD), are the leading indications for colon surgery in children. While these diseases have low mortality rates and surgical techniques can effectively restore anatomy, these patients have persistent and significant post-operative morbidity around fecal soiling and/or constipation. In addition to impairing growth and development, this affects all domains of health related quality of life (HRQoL). Patients, families, and healthcare providers of children with these diseases consistently report that bowel management strategies that prevent soiling comprise one of the most important areas for high quality outcomes research.

Engaging patients and families to take an active role in their healthcare leads to improved outcomes. Providing physicians and families with near real-time data on outcomes in children with similar medical conditions can allow families to form realistic expectations and take an active role in their child's health. It also provides physicians with near real-time feedback on patient-reported outcome measures to guide both conversations and recommendations for therapy at the point-of-care. A rapid learning healthcare system (RLHS) is a system that merges clinical research and clinical care. It is designed to collect data during routine patient care and then utilize the data to rapidly generate evidence to improve patient care, provide information to patients and families, and track quality measures.

The investigators created a RLHS that integrates pre-specified data elements and validated surveys within the clinical workflow in order to operationalize automated research data collection and integrate predictive analytics into the electronic health record (EHR). To date, we have over 800 patients enrolled in the colorectal RLHS. Patients, caregivers, and physicians can access data in order to make informed, shared decisions about care and align expectations about outcomes.

The primary and secondary objective of this trial are as follows:

Primary Objective: To assess the ability of a RLHS to improve healthcare satisfaction in pediatric patients with complex colorectal diseases.

Secondary Objective: To assess the ability of a RLHS to improve patient-centered outcomes in pediatric patients with complex colorectal diseases.To characterize the usability of the RLHS by patients and caregivers.

ELIGIBILITY:
Inclusion Criteria:

* English speaking patients aged 0-17 years with a diagnosis of ARM, HD, or functional constipation referred to our CCPR clinic between July 1, 2016 through June 1, 2017.

Exclusion Criteria:

* Patients previously treated at CCPR, those who are non-English speaking, and those without internet access.

Max Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 133 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Improved healthcare satisfaction | 30 days post-enrollment
  To assess the ability of a RLHS to improve healthcare satisfaction in pediatric patients with complex colorectal diseases. As measured by the PedsQL Healthcare Satisfaction questionnaire

SECONDARY OUTCOMES:
Improved patient-centered outcomes | 30 days post-enrollment
  To assess the ability of a RLHS to improve patient-centered outcomes in pediatric patients with complex colorectal diseases. As measured by the PedsQL Quality of Life questionnaire designed for both parents and children.
Usability of RLHS | 30 days post-enrollment
  To characterize the usability of the RLHS by patients and caregivers. As measured by the System Usability Scale designed by the investigators.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Deans, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No